CLINICAL TRIAL: NCT00656214
Title: Efficacy of Oral Lycopene in the Management of Oral Lichen Planus
Brief Title: Treatmant of Oral Lichen Planus With Lycopene
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: College of Dental Sciences, India (Other)
Responsible Party: College of Dental Sciences, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: olplycopene
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2004-11

CONDITIONS: Lichen Planus, Oral
Keywords: Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral; Lichen Planus | interventions — Lycopene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Active Comparator): Patients with symptomatic oral lichen planus
  Interventions: Drug: Lycopene
- B (Placebo Comparator): Patients with symptomatic oral lichen planus
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lycopene — 08 mg/day in two divided dosage
  Other Names: Lycored (Jagsonpal Pharmaceuticles, India)
  Arms: A
Drug: Placebo — Two divided dosage
  Arms: B

SUMMARY:
the purpose of this study was to evaluate that if lycopene, a potent antioxidant can be used in the treatment of oral lichen planus. this could be useful as lycopene has no reported side effects and hence it can used in place of steroids which are commonly used for this condition and have many reported adverse effects.

lycopene can be used in the treatment of this condition as free radicals have been found to play a role in the cause of this disease and also lower levels of lycopene were seen in these patints.

DETAILED DESCRIPTION:
Lichen planus, a chronic inflammatory mucocutaneous disease, occurs in about 2% of the adult population, affecting the skin and or oral mucosa. Clinically, lichen planus appears in keratotic, atrophic or erosive form. The atrophic and erosive forms are usually symptomatic.

Various treatment modalities viz. corticosteroids, antimicrobials, immunomodulators, phenytoin, retinoids, UV-radiation and surgical treatment etc. have been tried. Though none of these have shown to achieve satisfactory results with recurrence of lesion occurring in most of the cases after few weeks of discontinuation of therapy.

Recently a population based case control study has revealed lower levels of lycopene in atrophic and erosive oral lichen planus cases, while no significant difference was noted in any other carotenoid levels.

Lycopene is an antioxidant and free radical scavenger being used in the management of infertility, pre-eclampsia, cataract prevention, osteoarthritis, as adjuvant therapy in various malignancies, cardiovascular disorders, diabetes mellitus, aging, Alzheimer's disease, parkinsonism, etc.

Systemic lycopene has been found to be effective in treatment of oral leukoplakia, owing to its antioxidant properties.

The utility of lycopene in oral lichen planus has not been reported in the literature; therefore, this study has been designed to assess the efficacy of systemic lycopene in management of oral lichen planus patients.

The data collected from this study can move us closer to deriving a specific treatment plan for oral lichen planus - a dividend, not only for patients but dental fraternity as well.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were physically healthy and well oriented in time space and as a person.
2. Patients clinically & histopathologically diagnosed to be suffering from oral lichen planus.
3. Patients who had symptoms i.e. pain and/or burning sensation secondary to oral lichen planus.
4. Patients not on any treatment for the same. In case they were, then such treatment was stopped and a washout period of two weeks was given.
5. Patients who agreed to take medication supplied.
6. Patients who were willing for evaluation once in every two weeks for 8 weeks and also agreed to follow up every 30 days for 60 days.
7. Patients who agreed for the biopsy and hematological examination.

Exclusion Criteria:

1. Patients suffering from any systemic disease/s like Diabetes, Hypertension, Cardiovascular system disease, Renal dysfunction, Liver disorders etc.
2. Patients with any other mucosal disease or any other skin disease which may be associated with oral lesions.
3. Patients on any drug therapy which may cause lichen planus like lesions.
4. Patients with findings of any physical or mental abnormality, which would interfere with or be affected by the study procedure.
5. Patients with a known allergy or contraindication to study medications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Relief from signs & symptoms of disease | 08 weeks

SECONDARY OUTCOMES:
Relief from signs & symptoms of disease | 08 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dr MC Shashikanth, MDS, Study Director — Professor & Head of Department, Department of Oral Medicine & Radiology, College of Dental Sciences, Davangere, Karnataka, India
Locations (1):
- Department of oral medicine & radiology, College of dental sciences, Davangere, Karnataka, India

REFERENCES:
- [Background] Nagao T, Warnakulasuriya S, Ikeda N, Fukano H, Yamamoto S, Yano M, Miyazaki H, Ito Y. Serum antioxidant micronutrient levels in oral lichen planus. J Oral Pathol Med. 2001 May;30(5):264-7. doi: 10.1034/j.1600-0714.2001.300502.x. PMID 11334461
- [Background] Lycopene. Monograph. Altern Med Rev. 2003 Aug;8(3):336-42. No abstract available. PMID 12946243
- [Background] Singh M, Krishanappa R, Bagewadi A, Keluskar V. Efficacy of oral lycopene in the treatment of oral leukoplakia. Oral Oncol. 2004 Jul;40(6):591-6. doi: 10.1016/j.oraloncology.2003.12.011. PMID 15063387